CLINICAL TRIAL: NCT03818750
Title: Impact of Marketing of Alcohol Products on Young People
Acronym: IMAJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ecole des Hautes Etudes en Santé Publique (EHESP) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC18_8845_IMAJ; 2018-A00219-46 (Other: ID-RCB)
Record Dates: First submitted 2018-09-05; First posted 2019-01-28 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients (60) will be selected from the Alcohol Use Disorders Identification Test (AUDIT-C) :
  * "light drinkers" (score between 1 to 3)
  * "heavy drinkers" (score between 4 to 7) Two clinical visits will be realized in less than 4 weeks
  Interventions: Device: MRI; Behavioral: Alcohol Use Disorders Identification Test

INTERVENTIONS:
Device: MRI — Subjects review alcohol ads in different contexts (neutral context vs positive context such as parties and sport) and answer with buttons lever while being in the MRI to express their desire to consume alcohol or not.
  Subjects will be exposed to 288 ads set up.
Behavioral: Alcohol Use Disorders Identification Test — Questionnaire

SUMMARY:
Impact of marketing of alcohol products on young people

DETAILED DESCRIPTION:
Responsible for 3.3 million deaths worldwide, alcohol consumption causes diseases (liver cirrhosis, cancers, etc.) and social problems (injuries, road accidents, alcohol dependence, etc.). With one of the highest consumption rate in Europe, alcohol is the second cause of avoidable mortality in France after tobacco (49.000 alcohol attributable deaths in 2009) and its social cost is estimated to 120 billion euros. French teenage population is particularly associated with heavy drinking patterns: in 2014, 49% of 17-year olds declared heavy episodic drinking.

In that regard, several measures are recommended by health actors to combat this issue: minimum unit pricing, sales ban to minor, low blood alcohol concentration for drivers, etc. A specific measure concerns alcohol advertising restrictions. Some countries implemented alcohol advertising regulation laws (Poland, Sweden, Finland, Estonia, etc.), including France with the Evin law passed in 1991. This French law mandates advertising (and packaging) content to strictly convey factual information and objective qualities of alcohol products and thus bans attractive ads based on image and lifestyle evocations (seduction, power, etc.).

The objective of this research is to investigate whether statutory framework for alcohol advertising (e.g., Evin law) can effectively protect people against misleading, suggestive, and appealing content. Little research has been conducted on this topic in spite of WHO's recommendations (most research has explored the influence of exposure to ads but not the impact of content).

ELIGIBILITY:
Inclusion Criteria:

* volunteer males
* aged 18-25
* right-handed
* persons that consume alcohol : " light drinkers " or "heavy drinkers" (defined with the AUDIT scale, scores between 1 to 7)
* written consent and agreement consent will be given
* Affiliated to the French social insurance

Exclusion Criteria:

* color-blind persons
* misuse of psychoactive products (except tobacco) (cannabis : no regular consumers -more than 10 times per month ; no users of other illicit drugs - even for occasional consumption)
* non fluent french speaking persons (people who couldn't understand instructions or asked questions)
* persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Related to the MRI:

* Cardiac pacemaker or implanted defibrillator
* Cochlear implant
* Peripheral or neuronal stimulator
* Intra-ocular or brain metallic foreign bodies
* Any other contraindications to MRI

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Changes in brain activation in areas involved in the control of reward and motivation when looking at neutral versus contextual ads | Month 1
  Significant change in cerebral activity (expressed as a significant variation in hemodynamic response BOLD) in the condition of alcohol ads with versus without context (party, sport, people) in areas involved in the control of reward and motivation (striatum dorsal, insula)

CONTACTS AND LOCATIONS:
Overall Officials: Romain Moirand, MD, PhD, Principal Investigator — CHU of Rennes
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No